CLINICAL TRIAL: NCT00549835
Title: Acupuncture for Mucositis Pain in Cancer Care
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate funding
Sponsor: Johns Hopkins University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NA_00008179
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-03

CONDITIONS: Mucositis; Pain; Leukemia
Keywords: mucositis pain; cancer; pain; acupuncture; mucositis; cancer pain
MeSH Terms: conditions — Mucositis; Pain; Leukemia; Neoplasms; Cancer Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real Acupuncture (Active Comparator): Participants will have acupuncture performed at a rate of 3 times (Mon, Wed, Fri) / week for total of 2 weeks (total of 6 sessions). We will follow Saam Acupuncture methods, which have been the mainstream of acupuncture methodology in most Korean Oriental Medical Colleges and among clinical practitioners >400 years. Standardized acupuncture prescriptions for mucositis will be acupuncture points tonifying Spleen Meridian (R side) and Small Intestine Meridian (L side). In Oriental Medicine, the spleen has functions of promoting water metabolism, transporting nutrients, and controlling blood. Mouth belongs to the spleen system according to Five element theory. Small intestine is related with mucositis symptoms including thirst and tongue ulcers. We will use sterile, disposable, filiform needles, size 0.16 (40Gauge) - 0.30 mm (30Gauge) in diameter and 15-40 mm long. Total number of acupuncture needles will be 8 (4 needles each side) and needles will be retained for 20 minutes.
  Interventions: Procedure: Real Acupuncture; Procedure: Sham Acupuncture
- Sham Acupuncture (Sham Comparator): Newly diagnosed leukemia patients will be recruited from the large patient population on the Leukemia Inpatient Services who will be receiving high dose preperative regimens such as Busulfan + Cytarabine for marrow transplantation.
  Interventions: Procedure: Real Acupuncture; Procedure: Sham Acupuncture

INTERVENTIONS:
Procedure: Real Acupuncture
Procedure: Sham Acupuncture — Sham needles are developed to exclude sham effect and to prove real acupuncture efficacy. We will use specifically retractable Park Sham Device (AcuPrime, Exeter, UK) for control group. Because this sham device gives the impression of insertion with telescopic needle body and some pricking sensation with a bunt needle tip. It is a valid control for many acupuncture trials as it doesn't penetrate skin and doesn't create active stimulation as much as real needles or acupressure. To avoid unnecessary stimulation of penetrating skin in this population, we plan to use non-penetrating sham device rather than penetrating non-acupuncture point with real needles as control intervention.
  All other procedures will be same as Real Acupuncture group except using non-penetrating sham needles on non-acupuncture points. After final session, we will ask all subjects in both groups which form of treatment each subject believe to have during study and will analyze blinding credibility.

SUMMARY:
This research is being done to see if acupuncture helps relieve mucositis pain in patients with leukemia who are undergoing chemotherapy. Many patients receiving chemotherapy develop mucositis (painful sores or blisters in the mouth or throat). Mucositis is not only a frequent complication in cancer care and extremely painful, but also increases the risks of infection and malnutrition and often leads to discontinuing or delaying the chemotherapy treatments.

DETAILED DESCRIPTION:
Acupuncture is one of the oldest, most commonly used medical procedures in the world. The practice originated in China more than 2,000 years ago, and is widely used by doctors in Korea, China, Japan, and other countries to ease pain or various symptoms. In the past two decades, acupuncture has grown in popularity in the United States, and by 2002, an estimated 8.2 million adults in the US report having used acupuncture.

The term acupuncture describes a family of procedures involving stimulation of anatomical points on the body by a variety of techniques. The acupuncture technique that has been most studied scientifically involves penetrating the skin with thin, solid, metallic needles that are manipulated by the hands or by electrical stimulation. Acupuncture needles are metallic, solid, and hair-thin. People experience acupuncture differently, but most feel no or minimal pain as the needles are inserted. Some people are energized by treatment, while others feel relaxed.

Acupuncture has been used to ease some cancer treatment-related side effects such as nausea and vomiting. In this study we will assess the potential usefulness of acupuncture to ease the pain associated with mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with leukemia (such as acute myelogenous leukemia) and receiving chemotherapy for induction, consolidation or re-induction or high dose preparative regimen for bone marrow transplantation in the Johns Hopkins Oncology Inpatient Services
* Participation in standard leukemia-treatment regimens
* Expectation of survival of three weeks for completion of the study

Exclusion Criteria:

* Acupuncture treatment within the previous 6 weeks
* Unable to achieve platelet count of at least 10,000 with platelet support
* Radiation therapy within one month of enrollment
* Pregnant women
* History of substance abuse, including alcohol and IV drug users

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Compliance | 12 weeks
  Retention/ dropout rate
Sham credibility rate | 12 weeks
Frequency of any adverse effects | 12 weeks
  Bleeding, infection, bruising, etc

SECONDARY OUTCOMES:
Pain levels | 12 weeks
Mucositis Grade | 12 weeks
  CTC Scoring, Hopkins Scoring; Oral Mucositis Daily Questionnaire (OMDQ)
Total amount of conventional analgesics used and Total days on Analgesic | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adrian S Dobs, MD MHS, Principal Investigator — Johns Hopkins University; Sanghoon Lee, KMD PhD LAc, Study Director — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States